CLINICAL TRIAL: NCT05268081
Title: Virtual Specialist Conferences Between General Practitioners and Endocrinologists About Type 2.Diabetes: a Pragmatic Randomized Controlled Trial
Brief Title: Specialist Conferences Between General Practitioners and Endocrinologists
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Region MidtJylland Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-30-72-353-21
Record Dates: First submitted 2022-01-31; First posted 2022-03-07 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Specialist conferences; Virtual conferences; Family physician; Endocrinologist; Type 2-diabetes; Randomized Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Masking description of intervention status, i.e., outcomes assessor will not know who received the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual specialist conferences (Experimental): The group of general practices who participates in the virtual specialist conferences with endocrinologists.
  Interventions: Other: Virtual specialist conferences
- Standard of care (No Intervention): Receives the usual, standard practice.

INTERVENTIONS:
Other: Virtual specialist conferences — The intervention consists of four virtual conferences (45 min each in month 2, 5, 8 and 11) and an introductory webinar (90 min in month 1) to learn GPs about how to use the electronic "Diabetes Overview" to identify and manage patients with T2D. Each general practice is assigned to one specific endocrinologist they meet with throughout. The four virtual conferences are thematic: T2D and cardiovascular disease and heart failure, T2D and lipids, T2D and kidney disease and blood pressure, and T2D and a free topic selected by the GP. At each conference, the GP must bring 2-3 patient cases related to the theme and 1-2 patients of their own choice. The GP chairs the meeting. Each conference follows the same format: Check in (5 min); Short presentation by the endocrinologist (10 min); Presentation by GP and joint dialogue about theme-related patients (20 min); Presentation by GP and joint dialogue about theme-unrelated patients (optional, 5 min); (5) Wrapping-up (5 min).
  Arms: Virtual specialist conferences

SUMMARY:
To support the primary care sector in delivering high-quality Type 2-diabetes (T2D), literature reviews emphasize the need for implementing models of collaboration that in a simple and effective way facilitate clinical dialogue between general practitioners (GPs) and endocrinologists. The overall aim of the project is to study if an intervention consisting of structured cross-sectoral and virtual conferences between GPs and endocrinologists about T2D improves diabetes care and increases diabetes competencies and management in general practice. This aim will be studied in a pragmatic randomized controlled trial design. This potential is yet to be fully tapped because of methodological limitations. Studies have also not yet systematically evaluated virtual conferences in the context of chronic care using a high-quality research design.

DETAILED DESCRIPTION:
The overall aim is to study if cross-sectoral and virtual specialist conferences improves diabetes care and increases diabetes competencies and management in general practice. The expectation is that the intervention will:

at the patient level:

* improve adherence to international recommendations on diabetes medication for patients with Type 2-diabetes (T2D)
* improve the risk profile of patients with T2D with a reduction in glycated haemoglobin, blood pressure and cholesterol

at the general practice level:

- improve the self-reported competence and confidence in management of patients with T2D among general practitioners and practice staff

The intervention consists of four virtual and thematic conferences: (1) T2D and cardiovascular disease and heart failure, (2) T2D and lipids, (3) T2D and kidney disease and blood pressure, and (4) T2D and a free topic selected by the general practitioner (GP). Before having the first virtual conference, an introductory webinar is held to learn GPs about how to use the electronic "Diabetes Overview" to identify and manage patients with T2D. Each general practice is assigned to an endocrinologist who they meet at all four conferences. The intervention was developed using the Medical Research Framework for developing complex interventions.

All general practices located in the Municipality of Aarhus, Denmark are invited (n = 100). Block randomization is performed at the general practice level, and general practices will be randomized in a 1:1 ratio to either the intervention or the control group.

ELIGIBILITY:
Inclusion Criteria:

* General practices are eligible for inclusion if licensed and located in the municipality of Aarhus.
* GPs must consent to participate in the intervention and collect the data needed to measure patient and general practice outcomes.
* GPs must agree to bring patient cases to the virtual conferences who are ≥18 years, diagnosed with T2D and who they would like to discuss with the endocrinologist.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Ischemic heart disease and/or stroke treated with GLP1-RA and SGLT2 inhibitor | Month 12
  Percentage of patients with type 2-diabetes and ischemic heart disease and/or stroke being treated with glucagon-like peptide 1 receptor agonists (GLP1-RA) and sodium glucose cotransporter 2 (SGLT2) inhibitor
Micro/macro-albuminuria treated with ACE-inhibitor or AT2 | Month 12
  Percentage of patients with type 2-diabetes and micro/macro-albuminuria being treated with Angiotensin-converting-enzyme-inhibitor (ACE) or angiotensin-2-receptorantagonist (AT2)
LDL>2.5 mmol/L treated with Statins | Month 12
  Percentage of patients with type 2-diabetes and LDL>2.5 mmol/L being treated with Statins
Questionnaire for the assessment of general practitioners' confidence in managing type-2 diabetes in general | Month 12
  Self-reported degree to which the general practitioner is confident in: managing diabetes; managing patients with diabetes; managing patients with complex diabetes; managing patients with diabetes who are non-compliant.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of general practitioners' skills in managing type-2 diabetes in general | Month 12
  Self-reported degree to which the general practitioner is confident in: assessing when it is appropriate to initiate insulin treatment; selecting the appropriate medicine, when patients with diabetes need three-agent antidiabetics; selecting the appropriate medicine, when patients with have co-morbidity; achieving a lower level of Hb1Ac in patients with diabetes; high treatment quality for patients with diabetes; setting treatment targets for patients with diabetes; referring the right patients with diabetes to the department of endocrinology.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of general practitioners' confidence in managing type-2 diabetes and cardiovascular disease or heart failure | Month 12
  Self-reported degree to which the general practitioner is confident in: managing cardiovascular disease in patients with diabetes; assessing risk of cardiovascular disease in patients with diabetes; selecting the most appropriate medication for patients with diabetes and cardiovascular disease; achieving high treatment quality for patients with diabetes and cardiovascular disease; managing heart failure in patients with diabetes; assessing risk of heart failure in patients with diabetes; selecting the most appropriate medication for patients with diabetes and heart failure; achieving high treatment quality for patients with diabetes and heart failure.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of general practitioners' confidence in managing type-2 diabetes and blood pressure | Month 12
  Self-reported degree to which the general practitioner is confident in: managing high blood pressure in patients with diabetes; selecting the most appropriate medication for patients with diabetes and high blood pressure; achieving high treatment quality for patients with diabetes and high blood pressure.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of general practitioners' confidence in managing type-2 diabetes and kidney disease | Month 12
  Self-reported degree to which the general practitioner is confident in: managing kidney disease in patients with diabetes; managing Estimated Glomerular Filtration Rate (eGFR) in patients with diabetes; managing albuminuria in patients with diabetes; selecting the most appropriate medication for patients with diabetes if they have kidney disease in the form of lowered eGFR; selecting the most appropriate medication for patients with diabetes if they have kidney disease in the form of albuminuria; achieving high treatment quality for patients with diabetes and kidney disease.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of general practitioners' confidence in managing type-2 diabetes and cholesterol | Month 12
  Self-reported degree to which the general practitioner is confident in: managing high cholesterol in patients with diabetes; selecting the most appropriate cholesterol lowering medication for patients with diabetes; achieving a lower level of cholesterol among patients with diabetes and high cholesterol.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.

SECONDARY OUTCOMES:
Ischemic heart disease and/or stroke treated with GLP1-RA and SGLT2 inhibitor | Month 24
  Percentage of patients with type 2-diabetes and ischemic heart disease and/or stroke being treated with glucagon-like peptide 1 receptor agonists (GLP1-RA) and sodium glucose cotransporter 2 (SGLT2) inhibitor
Micro/macro-albuminuria treated with ACE-inhibitor or AT2 | Month 24
  Percentage of patients with type 2-diabetes and micro/macro-albuminuria being treated with Angiotensin-converting-enzyme-inhibitor (ACE) or angiotensin-2-receptorantagonist (AT2)
LDL>2.5 mmol/L treated with Statins | Month 24
  Percentage of patients with type 2-diabetes and LDL>2.5 mmol/L being treated with Statins
Questionnaire for the assessment of general practitioners' confidence in managing type-2 diabetes in general at 24 month | Month 24
  Self-reported degree to which the general practitioner is confident in: managing diabetes; managing patients with diabetes; managing patients with complex diabetes; managing patients with diabetes who are non-compliant.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of general practitioners' skills in managing type-2 diabetes in general at 24 month | Month 24
  Self-reported degree to which the general practitioner is confident in: assessing when it is appropriate to initiate insulin treatment; selecting the appropriate medicine, when patients with diabetes need three-agent antidiabetics; selecting the appropriate medicine, when patients with have co-morbidity; achieving a lower level of Hb1Ac in patients with diabetes; high treatment quality for patients with diabetes; setting treatment targets for patients with diabetes; referring the right patients with diabetes to the department of endocrinology.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of general practitioners' confidence in managing type-2 diabetes and cardiovascular disease or heart failure at 24 month | Month 24
  Self-reported degree to which the general practitioner is confident in: managing cardiovascular disease in patients with diabetes; assessing risk of cardiovascular disease in patients with diabetes; selecting the most appropriate medication for patients with diabetes and cardiovascular disease; achieving high treatment quality for patients with diabetes and cardiovascular disease; managing heart failure in patients with diabetes; assessing risk of heart failure in patients with diabetes; selecting the most appropriate medication for patients with diabetes and heart failure; achieving high treatment quality for patients with diabetes and heart failure.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of general practitioners' confidence in managing type-2 diabetes and blood pressure at 24 month | Month 24
  Self-reported degree to which the general practitioner is confident in: managing high blood pressure in patients with diabetes; selecting the most appropriate medication for patients with diabetes and high blood pressure; achieving high treatment quality for patients with diabetes and high blood pressure.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of general practitioners' confidence in managing type-2 diabetes and kidney disease at 24 month | Month 24
  Self-reported degree to which the general practitioner is confident in: managing kidney disease in patients with diabetes; managing Estimated Glomerular Filtration Rate (eGFR) in patients with diabetes; managing albuminuria in patients with diabetes; selecting the most appropriate medication for patients with diabetes if they have kidney disease in the form of lowered eGFR; selecting the most appropriate medication for patients with diabetes if they have kidney disease in the form of albuminuria; achieving high treatment quality for patients with diabetes and kidney disease.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of general practitioners' confidence in managing type-2 diabetes and cholesterol at 24 month | Month 24
  Self-reported degree to which the general practitioner is confident in: managing high cholesterol in patients with diabetes; selecting the most appropriate cholesterol lowering medication for patients with diabetes; achieving a lower level of cholesterol among patients with diabetes and high cholesterol.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Patients with T2D and HbA1c <58 mmol/L at 12 and 24 months | Month 12 and Month 24
  Percentage of patients with type 2-diabetes and HbA1c <58 mmol/L
Patients with T2D and HbA1c <53 mmol/L at 12 and 24 months | Month 12 and Month 24
  Percentage of patients with type 2-diabetes and HbA1c <53 mmol/L
Patients with T2D and blood pressure <140 mmHg at 12 and 24 months | Month 12 and Month 24
  Percentage of patients with type 2-diabetes and blood pressure <140 mmHg
Patients with T2D and blood pressure <130 mmHg at 12 and 24 months | Month 12 and Month 24
  Percentage of patients with type 2-diabetes and blood pressure <130 mmHg
Patients with T2D and LDL >2.5 mmol/L at 12 and 24 months | Month 12 and Month 24
  Percentage of patients with type 2-diabetes and low-density lipoprotein >2.5 mmol/L
Patients with T2D and microalbuminuria and LDL >1.8 mmol/L at 12 and 24 months | Month 12 and Month 24
  Percentage of patients with type 2-diabetes and microalbuminuria and LDL >1.8 mmol/L
Questionnaire for the assessment of general practitioners' rating of relational coordination in the general practice at 12 and 24 months | Month 12 and Month 24
  Self-reported assessment by the general practitioner about their collaboration with the general practice using the relational coordination survey that measures the degree of: Frequent Communication; Timely Communication; Accurate Communication; Problem Solving Communication; Shared Goals; Shared Knowledge; Mutual Respect.
  Range 1-5, higher score indicates relational coordination.
Questionnaire for the assessment of general practitioners' rating of relational coordination with the hospital at 12 and 24 months | Month 12 and Month 24
  Self-reported assessment by the general practitioner about their collaboration with the hospital using the relational coordination survey that measures the degree of: Frequent Communication; Timely Communication; Accurate Communication; Problem Solving Communication; Shared Goals; Shared Knowledge; Mutual Respect.
  Range 1-5, higher score indicates relational coordination.
Questionnaire for the assessment of general practitioners' rating of using virtual conferences at 12 and 24 months | Month 12 and Month 24
  Self-reported assessment by the general practitioner about using virtual conferences measured along the four dimensions of the Technology Acceptance Model: perceived usefulness of virtual conferences; perceived ease-of-use of virtual conferences; attitude to using virtual conferences; behavioural intention as regards using virtual conferences.
  Range 1-5 from "completely disagree" to "completely agree", higher score indicates higher user ratings.
Questionnaire for the assessment of practice staffs' rating of relational coordination in the general practice at 12 and 24 months | Month 12 and Month 24
  Self-reported assessment by the practice staff about their collaboration with the general practice using the relational coordination survey that measures the degree of: Frequent Communication; Timely Communication; Accurate Communication; Problem Solving Communication; Shared Goals; Shared Knowledge; Mutual Respect.
  Range 1-5, higher score indicates higher relational coordination.
Questionnaire for the assessment of practice staffs' rating of relational coordination with the hospital at 12 and 24 months | Month 12 and Month 24
  Self-reported assessment by the practice staff about their collaboration with the hospital using the relational coordination survey that measures the degree of: Frequent Communication; Timely Communication; Accurate Communication; Problem Solving Communication; Shared Goals; Shared Knowledge; Mutual Respect.
  Range 1-5, higher score indicates higher relational coordination.
Questionnaire for the assessment of practice staffs' rating of using virtual conferences at 12 and 24 months | Month 12 and Month 24
  Self-reported assessment by the practice staff about using virtual conferences measured along four dimensions of the Technology Acceptance Model: perceived usefulness of virtual conferences; perceived ease-of-use of virtual conferences; attitude to using virtual conferences; behavioural intention as regards using virtual conferences.
  Range 1-5 from "completely disagree" to "completely agree", higher score indicates higher user ratings.
Questionnaire for the assessment of practice staffs' confidence in managing type-2 diabetes in general at 12 and 24 month | Month 12 and Month 24
  Self-reported degree to which the practice staff is confident in: managing diabetes; managing patients with diabetes; managing patients with complex diabetes; managing patients with diabetes who are non-compliant; achieving high treatment quality for patients with diabetes.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of practice staffs' confidence in managing type-2 diabetes and cardiovascular disease or heart failure at 12 and 24 month | Month 12 and Month 24
  Self-reported degree to which the practice staff is confident in: managing cardiovascular disease in patients with diabetes; assessing risk of cardiovascular disease in patients with diabetes; achieving high treatment quality for patients with diabetes and cardiovascular disease; managing heart failure in patients with diabetes; assessing risk of heart failure in patients with diabetes; achieving high treatment quality for patients with diabetes and heart failure.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of practice staffs' confidence in managing type-2 diabetes and blood pressure at 12 and 24 months | Month 12 and Month 24
  Self-reported degree to which the practice staff is confident in: managing high blood pressure in patients with diabetes; achieving high treatment quality for patients with diabetes and high blood pressure.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of practice staffs' confidence in managing type-2 diabetes and kidney disease at 12 and 24 months | Month 12 and Month 24
  Self-reported degree to which the practice staff is confident in: managing kidney disease in patients with diabetes; achieving high treatment quality for patients with diabetes and kidney disease.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.
Questionnaire for the assessment of practice staffs' confidence in managing type-2 diabetes and cholesterol at 12 and 24 month | Month 12 and Month 24
  Self-reported degree to which the practice staff is confident in managing high cholesterol in patients with diabetes.
  Range 1-5 from "not at all" to "a very high degree", higher score indicates higher confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Thim Prætorius, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus N, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Restrictions apply to the availability of these datasets. Register data will be used under license for the current study. Survey data and patient outcomes data are not publicly available as per the written consent signed by general practitioners and endocrinologists. Data are, however, available for research purposes from the authors upon reasonable request and with permission from study participants.

REFERENCES:
- [Background] Praetorius T, Baymler Lundberg AS, Sondergaard E, Tang Knudsen S, Sandbaek A. The effect of virtual specialist conferences between endocrinologists and general practitioners about type 2 diabetes: study protocol for a pragmatic randomized superiority trial. Trials. 2022 Dec 28;23(1):1059. doi: 10.1186/s13063-022-06961-y. PMID 36578024
- [Derived] Praetorius T, Baymler Lundberg AS, Klausen Fredslund E, Blach Rossen N, Gregersen S, Prior A, Sondergaard E, Tang Knudsen S, Sandbaek A. Effect of video conferencing between primary and secondary care specialists on type 2 diabetes medication. NPJ Digit Med. 2025 Mar 28;8(1):179. doi: 10.1038/s41746-025-01570-w. PMID 40148532
- See also: Related Info — https://www.stenoaarhus.dk/forskning/deltag-i-forskningsprojekter/star/